CLINICAL TRIAL: NCT06659601
Title: Deep Learning Model to Predict the Recurrence of Stage IA Invasive Lung Adenocarcinoma After Sub-lobar Resection
Acronym: DL-Rec-ILA
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xin Fan, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2022MSXM147; 2022MSXM147 (Other Grant/Funding Number: Joint project of Chongqing Health Commission and Science and Technology Bureau)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Focus on Developing a Deep Learning Model to Predict the Recurrence Risk of Stage IA Invasive Lung Adenocarcinoma After Sub-lobar Resection
Keywords: Lung cancer; Sub-lobar resection; Computed tomography; Deep learning
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Training Cohort: Patients in this cohort diagnosed with stage IA invasive lung adenocarcinoma who underwent sub-lobar resection. This cohort is used to train the 3D deep learning model to predict recurrence risk.
- Validation Cohort: Patients in this cohort with stage IA ILADC. It is used to validate the model performance internally and assess its generalization within the same institution。
- Testing Cohort: Patients in this cohort from other institution. It is used to test the generalizability of the model in predicting recurrence risk in an independent dataset.

SUMMARY:
This study aims to develop a deep learning model based on noncontrast CT images to predict the recurrence risk of stage IA invasive lung adenocarcinoma after sub-lobar resection，which can serve as potential tool to assist thoracic surgeons in making optimal treatment decisions.The study will use existing CT data to train and validate the model, without requiring any additional intervention for the participants.

DETAILED DESCRIPTION:
This study is designed to develop a deep learning model to predict the recurrence risk of stage IA invasive lung adenocarcinoma after sub-lobar resection using noncontrast CT images. The best indications for sub-lobar resection in patients with early-stage LADC are still debated, making surgical method selection somewhat difficult. The deep learning model can noninvasively and objectively predict the recurrence risk of patients with stage IA ILADC following sub-lobectomy and are helpful in predicting prognosis of patients with stage IA ILADC after sub-lobectomy and can facilitate the choosing of the optimal surgery mode of these patients.

The study will utilize retrospective data from patients with stage IA invasive lung adenocarcinoma after sub-lobar resection . Noncontrast CT images will be collected at admission and used as inputs for the deep learning model. The model will be trained using convolutional neural networks (CNN) to identify patterns associated with recurrence.

In addition to model development, the study will also evaluate the model's performance on a separate validation cohort to assess generalizability. Statistical analyses will include performance metrics such as area under the receiver operating characteristic (ROC) curve (AUC) and precision-recall curve.

This study aims to provide a valuable tool for clinicians to make timely decisions in choosing the optimal therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:(i) pathological confirmation of LADC; (ii) undergoing sub-lobar resection (wedge resection or segmentectomy); (iii) CT scanning prior to surgery; (iv) pathological staging of IA; and (v) complete clinical and follow-up data.

-

Exclusion Criteria:(i) multiple primary LADC; and (ii) other pulmonary lesions that might interfere with the morphological assessment of tumors.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients diagnosed with stage IA invasive lung adenocarcinoma (ILADC) who underwent preoperative chest CT scans and sub-lobar resection. The participants are not limited in age, include both males and females, and were treated at our institution. The patients of external testing cohort are from other institution.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Recurrence Prediction Accuracy | October 2024
  The primary outcome measure is the accuracy of the 3D deep learning model in predicting the recurrence of stage IA invasive lung adenocarcinoma after sub-lobar resection. Accuracy will be evaluated by comparing the model's predictions with actual patient outcomes using metrics such as sensitivity, specificity, and area under the ROC curve (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Yuzhong District, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns and institutional regulations, individual participant data (IPD) will not be shared with external researchers.